CLINICAL TRIAL: NCT00103493
Title: Efficacy of a Tailored Oral Health Education Program
Brief Title: Oral Health Education Program
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Temple University (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); University of Michigan (Other); Delta Dental Fund of Michigan (Other)
Responsible Party: Amid Ismail, Principal Investigator, Temple University
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: NIDCR-14261; U54DE014261 (NIH)
Record Dates: First submitted 2005-02-09; First posted 2005-02-10 (Estimated); Last update posted 2010-11-22 (Estimated); Status verified 2009-07

CONDITIONS: Dental Caries; Oral Hygiene; Oral Health; Dental Health
MeSH Terms: conditions — Dental Caries | interventions — Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational interviewing
Behavioral: Targeted DVD-based educational program

SUMMARY:
The purpose of this study is to evaluate whether an oral health education program that is tailored to caregivers' understanding and acceptance of information on how to prevent tooth decay will lead to improvement in behaviors conducive to good oral health and reduction in tooth decay in his or her children.

DETAILED DESCRIPTION:
The Detroit Dental Health Project (DDHP) is a seven-year research study designed to identify the determinants of variation in prevalence and incidence of dental caries among low-income African-American children in Detroit. The children were randomly selected from housing units located in the lowest income areas (less than 250% of the poverty line). After over a year of preparation and testing, the DDHP listed over 18,000 housing and non-housing units in 118 randomly selected low-income neighborhoods in Detroit. A total of 12,000 housing units were randomly sampled and contacted over a period of one year (September 2001 - August 2002) in order to recruit a representative sample of African American children. Field interviewers contacted the selected housing units. The recruitment process located and scheduled around 1,400 families to visit the Dental Assessment Center (DAC). Of those, 1,021 visited the DAC and completed examinations and interviews (Phase I).

The long-term objective of this project is to develop an effective multi-component tailored/targeted behavioral intervention to promote and maintain good oral health and prevent oral diseases among low-income children. To achieve this, a multimedia-based multi-level intervention has been designed to be easy to use and easy to disseminate for large-scale use.

The efficacy of the Multi-Component Tailored/Targeted Intervention that will be delivered using motivational interviewing and a targeted educational video designed and produced for the specific population in comparison with the non-tailored health education (targeted educational video only - control group) will be tested in a randomized controlled trial. In Phase II of the Detroit Dental Health Project, the 1,021 low-income African Americans recruited will be randomly assigned to one of the two intervention groups. A dental examination will provide the baseline measurement and changes in the outcomes will be assessed in the follow-up examination after two years. Participants in the control and intervention groups will complete a questionnaire about their oral health and related behaviors. Participants in the control group will receive standard oral hygiene and caries risk counseling using only the educational video without any motivational interviewing (equivalent to a counseling session conducted by a dentist).

The 1,021 families have been randomized using a list of randomly generated numbers. The allocation of the assignment is being concealed from the analysis team and the examining dentist. After each session, the participants receive a "recipe" for oral health with a picture of their child. The control group participants receive a standard plan; whereas the caregivers in the intervention group receive the specific plan they have developed with the motivational interviewer.

After the intervention/control session, the participants are being followed by telephone contact to review the progress in oral health behaviors and answer questions. Follow-up questionnaires will be administered after 2-4 weeks, at 6 months, and 2 years after the intervention/control session.

ELIGIBILITY:
Inclusion Criteria:

* All participants have been randomly selected from 39 Census Tracts (CTs) in the city of Detroit. The tracts were selected based on household income using 2000 Census Data.
* Participants should live in one of the randomly selected dwellings in the selected CTs; have a child or children less than 6 years old at the time of recruitment in 2002-2003; and have a total family income of less than 250% percentile of the federal poverty line.

Exclusion Criteria:

* No family who is eligible was excluded from this study.

Ages: 15 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1021 (Actual)
Dates: Start 2004-10; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amid Ismail, Principal Investigator — University of Michigan
Locations (1):
- Dental Assessment Center, Detroit, Michigan, United States